CLINICAL TRIAL: NCT00779597
Title: Improvement of Self Management Skills for Oncologic Patients With Pain Through a Trans Institutional Nursing Intervention: a Cluster Randomized Multi Center Study
Brief Title: Improvement of Self Management for Oncologic Patients With Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Margarete Landenberger, Professor, Dr. phil. habil., Martin-Luther-University Halle-Wittenberg Medical Faculty, Department for Health and Nursing Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BMBF-T3; Grand No.: 01GT0601
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-10

CONDITIONS: Pain; Cancer
Keywords: self care; symptom management; pain; cancer; nurse coaching; patient education
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care as usual (No Intervention): Care as usual, i.e. standard pain treatment and standard care
- SCION-PAIN program (Experimental): SCION-PAIN program - Additionally to standard pain treatment, patients from the intervention wards received, the SCION-PAIN program consisting of 3 modules: pharmacologic pain management, non-pharmacologic pain management and discharge management.
  Interventions: Behavioral: SCION (Self care improvement through oncology nursing)-PAIN program

INTERVENTIONS:
Behavioral: SCION (Self care improvement through oncology nursing)-PAIN program — The intervention will be conducted by specially trained oncology nurses and will include the components of knowledge, skills training, and coaching to improve self care regarding pain management beginning with admission followed by booster session every third day and one follow up telephone counseling within 3 to 4 days after discharge from hospital.
  Arms: SCION-PAIN program

SUMMARY:
This study will test the SCION (Self care improvement through oncology nursing)-PAIN program, a multi-modular structured intervention to improve self management in oncologic patients with pain compared to care as usual (standard pain treatment and standard care). The study will determine if the self management skills of the patients continue to be used when the intervention stops, e.g. after discharge from hospital.

It is hypothesized that patients who receive the multi-modular structured intervention will have less patient-related barriers to the management of cancer pain.

DETAILED DESCRIPTION:
According to modified "Precede Model of health behavior" from Green, patients self management skills are affected by the patients' knowledge, activities and attitude to pain management.

Therefore, we conduct a cluster randomized clinical trial (C-RCT) that will test the effectiveness of SCION-PAIN program against care as usual on self pain management of the patient and average pain level.

As allocation to intervention or control is performed on the level of wards, randomization is stratified by ward profile (e.g. gynaecological, haematological, urological).

Wards were included if they agreed to participate and had more than 10% patients with a diagnosis of cancer in 2006. Wards with a pediatric profile were excluded.

Adult oncology patients with persistent pain will be recruited by the nurses of the participating wards under the guidance of a research nurse. Patients are included in the trial if they meet the inclusion criteria and sign informed consent. They will receive the intervention that the respective ward was allocated to.

The SCION-PAIN program as a multi modular structured nursing intervention (see Arm Description) will be conducted by specially trained ward nurses in cooperation with the research nurse. The intervention will include components of knowledge, skills training, and coaching (particularly against patient-related barriers to pain medication) to improve cancer pain management. Patients in intervention group will receive follow-up telephone counseling within 2 to 3 days after discharge. The self management skills of the patients will be observed up to 28 days post discharge. Both quantitative and qualitative analyses will be conducted to evaluate patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult oncology patients
* able to read, write, and understand German
* agree to participate and give informed consent
* have an average pain intensity score of > 3.0 on a 0 to 10 NRS
* pain persists for more than 3 days
* scheduled for another visit to the clinic

Exclusion Criteria:

* documented actual alcohol or drug abuse
* surgery within the last 3 days
* disorientated to date, place and situation
* have a ECOG Performance Score of 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Patient-related barriers to management of cancer pain (Barriers Questionnaire II) | 7 days after discharge

SECONDARY OUTCOMES:
Average pain intensity score (Brief Pain Inventory) | 7th day after discharge
HRQoL (EORTC QLQ C 30 (Version 3.0)) | 7th day after discharge
Adherence to pain medication (MORISKY Adherence Score) | 7th day after discharge
Coping of Pain (FESV-BW) | 7th day after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Margarete Landenberger, Professor, Dr., Principal Investigator — Martin-Luther-University Halle-Wittenberg; Ingrid Horn, Study Chair — University Hospital Halle, Martin-Luther-University Halle-Wittenberg; Anette Thoke-Colberg, Study Chair — University Hospital rechts der Isar, Munich Technical University
Locations (3):
- Germany (3):
  - University Hospital rechts der Isar, Munich Technical University, Munich, Bavaria
  - Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt
  - University Hospital Halle, Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt

REFERENCES:
- [Background] Jahn P, Kitzmantel M, Renz P, Kukk E, Kuss O, Thoke-Colberg A, Horn I, Landenberger M. Improvement of pain related self management for oncologic patients through a trans institutional modular nursing intervention: protocol of a cluster randomized multicenter trial. Trials. 2010 Mar 22;11:29. doi: 10.1186/1745-6215-11-29. PMID 20307262
- See also: Trial Protocol — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2855560/pdf/1745-6215-11-29.pdf